CLINICAL TRIAL: NCT05564143
Title: Endoscopic Ultrasound-guided Versus Surgical Gastroenterostomy for Malignant Gastric Outlet Obstruction: A Multi-centered Prospective Randomized Controlled Trial (ENCOURAGE Trial)
Brief Title: Endoscopic Ultrasound-guided Versus Surgical Gastroenterostomy for Malignant Gastric Outlet Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202204110RIPA
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-05

CONDITIONS: Malignant Gastric Outlet Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EUS-guided gastroenterostomy (EUS-GE) (Active Comparator): All EUS-GE procedures were performed under general anesthesia with endotracheal intubation. A forward-viewing gastroscope or side-viewing duodenoscope is first inserted into the site of the obstruction and a 0.025- or 0.035-inch stiff GW is placed down-stream of the jejunum beyond the obstruction as far as possible. Then, oral enteral tube is placed where the jejunum intended for stent placement under fluoroscopic guidance. After exchanging to EUS endoscope, the target jejunum is visualized by EUS after continuously injection of mixed saline and contrast medium. Finally, the gastrojejunostomy stent is directly advanced from the gastric wall into the target jejunum by AXIOS-EC delivery system.
  Interventions: Procedure: EUS-guided gastroenterostomy (EUS-GE)
- Laparoscopic gastroenterostomy (LGE) (Active Comparator): All LGE were performed in the operation room with patients under general anesthesia. After CO2 insufflation, 4 to 5 trocars were introduced. Next, the Treitz ligament was identified. An anterior, dorsal laterolateral, or side- to-side isoperistaltic gastroenteric anastomosis was constructed. The exact location of the gastroenteric anastomosis, with regard to the Treitz ligament, varied from 30 to 60 cm.
  Interventions: Procedure: Laparoscopic gastroenterostomy (LGE)

INTERVENTIONS:
Procedure: EUS-guided gastroenterostomy (EUS-GE) — Treatment
  Arms: EUS-guided gastroenterostomy (EUS-GE)
Procedure: Laparoscopic gastroenterostomy (LGE) — Treatment
  Arms: Laparoscopic gastroenterostomy (LGE)

SUMMARY:
Gastric outlet obstruction (GOO), defined by a mechanical obstruction of the duodenum, pylorus, or antrum, may result from various diseases. GOO was caused by underlying malignancy in up to 85% of patients, most of which could be attributed to pancreatic cancer. Malignant GOO may increase morbidity, reducing quality of life, and significantly influencing tolerability and efficacy of oncologic treatments. Before the advent of EUS-guided gastroenterostomy (EUS-GE), placement of enteral self-expandable metallic stents (SEMS) or surgical gastroenterostomy (SGE) are the standard of care for many years. The main shortcoming of enteral SEMS placement is recurrent GOO due to tumor ingrowth/overgrowth, which occurs in the majority of patients who survive longer than 6 months. On the other hand, the main limitation of SGE is its invasive nature, especially in such patients with advanced malignancies and poor nutritional status. In addition, SGE is associated with frequent complications, such as perioperative infections and gastroparesis.

EUS-guided gastroenterostomy (EUS-GE) is a novel procedure for palliation of malignant GOO. Several systematic reviews and meta-analysis demonstrated the feasibility, efficacy and safety of EUS-GE. Compared with laparoscopic GE (LGE), EUS-GE not only had almost identical technical and clinical success but also reduced time to oral intake, shorter median hospital stay, and lower rate of adverse events. However, data directly comparing EUS-GE to LGE are limited. We aimed to compare clinical outcomes between EUS-GE and LGE in the palliation of malignant GOO under a randomized setting.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients ≥ 20 years old
2. Confirmed unresectable distal gastric or duodenal or pancreatico-biliary malignancies
3. Suffering from gastric outlet obstruction with a gastric outlet obstruction score of ≤ 1
4. Performance status ECOG ≤3

Exclusion Criteria:

1. Unable to give informed consent
2. Prior duodenal metallic stent placement
3. Severe comorbidities precluding the endoscopic procedure or operation
4. Life expectancy of less than 1 month
5. History of gastric surgery
6. Linitus plastic
7. Multiple-level bowel obstruction confirmed on radiographic studies such as small bowel series or abdominal computed tomography
8. Coagulation disorders
9. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to functional recovery (days) | 1 week
  Functional recovery is reached when all of the following criteria are met: 1) adequate pain control with oral analgesia only, 2) restoration of mobility to an independent level (or to preoperative level if previously impaired, 3) ability to maintain sufficient caloric intake (minimum of 50% required calories), 4) absence of intravenous fluid administration, and 5) no signs of active abdominal infection.

SECONDARY OUTCOMES:
Technical success rate | 1 day
  The successful gastroenterostomy was confirmed by endoscopy or operation
Clinical success rate | 1 week
  Clinical success if measured by the improvement of at least 1 point in the gastric outlet obstruction score within one week after gastroenterostomy
Re-intervention rate | 6 months
  The percentage of patients requiring additional endoscopic intervention due to stent dysfunction
Duration of gastroenterostomy patency | 6 months
  Calculated from the time of gastroenterostomy creation to the time of gastroenterostomy dysfunction
Adverse events rates | 6 months
  Graded according to the lexicon of endoscopic adverse events
Gastric outlet obstruction scores (GOOS) | 6 months
  Scoring system for food intake. Range of score is 0 -3 with 3 being the highest and indicating tolerating full diet
Quality of life assessment scores | 6 months
  EORTC QLQ-C30. This questionnaire is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of 5 multiitem scales (physical, role, social, emotional and cognitive functioning) and 9 single items (pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life assessment scores | 6 months
  EORTC STO-22 modules. This the gastric cancer module to the QLQ-C30 questionnaire. The questionnaire is composed of 5 multiitem scales (dysphagia, pain, reflux, eating, anxiety) and 4 single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available